CLINICAL TRIAL: NCT06471725
Title: Effectiveness of Adding Pilates Exercises to Sports Hernia Rehabilitation:a Comparative Clinical Trial
Acronym: PESHR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohamed Ibrahim Elgohary, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F.P.T 2307016
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Pilates Exercises; Sports Hernia
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: 2X2 model
Who Masked: Participant, Outcomes Assessor
Masking Description: This study is a controlled, double-blinded (patients and assessors)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): will receive a combination of pilates exercises, Low-level laser therapy, and low-intensity ultrasound.
  Interventions: Other: combination of pilates exercises, Low-level laser therapy, and low-intensity ultrasound
- Control (Active Comparator): will be given Low-level laser therapy and low-intensity ultrasound
  Interventions: Other: combination of pilates exercises, Low-level laser therapy, and low-intensity ultrasound

INTERVENTIONS:
Other: combination of pilates exercises, Low-level laser therapy, and low-intensity ultrasound — The core and hip muscles will be targeted through a customized workout program consisting of exercises such as Breathing, Planks, Side- Planks, Weighted lunges, Glute Bridge, Clamshell, Half-Kneeling Hip Flexor Stretch, Swan dive, Roll down, Ab curls, and Shoulder bridge, Low-intensity Ultrasound , and low level laser therapy

SUMMARY:
The study recruited male sports hernias patients referred for physical therapy by an orthopedist or general practitioner from Damietta General Hospital. Participants had to be between 18 and 45 years old, have had sports hernia for two to ten weeks, and be willing and able to attend and stick to the Pilates exercise program for the trial's entire duration

DETAILED DESCRIPTION:
The study recruited male sports hernias patients referred for physical therapy by an orthopedist or general practitioner from Damietta General Hospital. Participants had to be between 18 and 45 years old, have had sports hernias for two to ten weeks, and be willing and able to attend and stick to the Pilates exercise program for the entire trial. Exclusion criteria were applied to patients with preexisting injuries or conditions that could affect Pilates exercise participation and those with contraindications or exacerbating conditions from such exercises. Further criteria were currently participating in other intensive exercise or rehabilitation programs and inability to give informed consent due to cognitive or communicative issues

ELIGIBILITY:
Inclusion Criteria:

* Participants had to be between 18 and 45 years old,
* have had sports hernia for two to ten weeks
* be willing and able to attend and stick to the Pilates exercise program for the trial's entire duration

Exclusion Criteria:

* patients with preexisting injuries or conditions that could affect Pilates exercise participation
* those with contraindications or exacerbating conditions from such exercises.
* currently participating in other intensive exercise or rehabilitation programs
* inability to give informed consent due to cognitive or communicative issues.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-06-19 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 12 weeks
  Typically, it consists of a 10 cm horizontal or vertical line with no pain at one end and the highest pain level at the other end.

SECONDARY OUTCOMES:
Lower Extremity Functional Scale | 12 weeks
  Consists of 20 items that assess the ability to perform activities related to lower extremity function, such as standing, walking, stair climbing, and balance.
Harris Hip Score | 12 weeks
  this tool is used to evaluate patients with hip conditions such as femoral neck fracture or OA.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Delta university for science and technology, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elabd OM, Etoom M, Jahan AM, Elabd AM, Khedr AM, Elgohary HM. The Efficacy of Muscle Energy and Mulligan Mobilization Techniques for the Upper Extremities and Posture after Breast Cancer Surgery with Axillary Dissection: A Randomized Controlled Trial. J Clin Med. 2024 Feb 8;13(4):980. doi: 10.3390/jcm13040980. PMID 38398293